CLINICAL TRIAL: NCT00157105
Title: Recombinant Antihemophilic Factor (rAHF PFM) Manufactured and Formulated Without Added Human or Animal Proteins: Evaluation of Safety and Efficacy in Hemophilia A Patients Undergoing Surgical or Invasive Procedures
Brief Title: Safety and Efficacy Study of a Recombinant and Protein-Free Factor VIII (rAHF-PFM) in Hemophilia A Patients Undergoing Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 069902
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

INTERVENTIONS:
Drug: Antihemophilic factor, recombinant, manufactured protein-free

SUMMARY:
The purpose of this study is to evaluate whether rAHF-PFM is safe and effective in the treatment of hemophilia A patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 5 years
* The subject has severe or moderately severe hemophilia A defined by a baseline factor VIII level <= 2% of normal documented at screening or historically (e.g., at hemophilia diagnosis)
* Subjects may enroll regardless of their serologic status for human immunodeficiency virus (HIV-1) and hepatitis C virus (HCV)
* The subject requires a surgical, dental or other invasive procedure--either elective or emergency
* The subject has a history of at least 150 exposure days for all other factor VIII products (as estimated by the study site investigator) prior to study entry
* The subject has a life expectancy of at least 28 days from the day of surgery
* The subject has been informed of the nature of the study, agreed to its provisions, and signed and dated the informed consent form approved by the appropriate IRB/IEC and Baxter BioScience

Exclusion Criteria:

* The subject has a detectable inhibitor to factor VIII in the local hemostasis laboratory at the investigative site at the time of enrollment
* The subject has a history of inhibitor to factor VIII > 1.0 BU. Note: If the subject has a history of an inhibitor titer > 1.0 BU at any time prior to enrollment but demonstrated expected clinical responses to conventional doses of factor VIII therapy, the subject may enroll
* The subject has known hypersensitivity to Recombinate
* The subject is currently participating in another investigational drug study, or has participated in any clinical trial involving an investigational drug within 30 days of study entry
* The subject has clinical and/or laboratory evidence of abnormal hemostasis from causes other than hemophilia A (e.g., late-stage chronic liver disease, immune thrombocytopenic purpura, disseminated intravascular coagulation)
* The subject is identified by the investigator as being unable or unwilling to cooperate with study procedures.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2001-02-12 (Actual); Primary Completion 2004-08-03 (Actual); Study Completion 2004-08-03 (Actual)

PRIMARY OUTCOMES:
Percent of participants experiencing treatment-related adverse experiences (AEs) | Throughout the study period of approximately 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- United States (10):
  - Children´s Hospital Los Angeles, Hemophilia Comprehensive Care Center, Division of Pediatric Hematology/Oncology, Los Angeles, California
  - Children´s Healthcare of Atlanta Blood Bank, Atlanta, Georgia
  - Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa Regional Hemophilia Center, Department of Pediatrics, Iowa City, Iowa
  - Brigham and Women´s Hospital, Hematology Division, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Mt. Sinai Medical School, Hemophilia Comprehensive Care Center, New York, New York
  - Children´s Hospital Medical Center Pharmacy, Hemophilia Treatment Center, Cincinnati, Ohio
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Puget Sound Blood Center, Seattle, Washington

REFERENCES:
- [Derived] Shapiro A, Gruppo R, Pabinger I, Collins PW, Hay CR, Schroth P, Casey K, Patrone L, Ehrlich H, Ewenstein BM. Integrated analysis of safety and efficacy of a plasma- and albumin-free recombinant factor VIII (rAHF-PFM) from six clinical studies in patients with hemophilia A. Expert Opin Biol Ther. 2009 Mar;9(3):273-83. doi: 10.1517/14712590902729392. PMID 19216617